CLINICAL TRIAL: NCT03541057
Title: Vienna Vascular Liver Disease Study: Characterization of Patients With Vascular Liver Disease - a Registry With Biobank
Brief Title: Vienna Vascular Liver Disease Study
Acronym: VALID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Thomas Reiberger, Assoc.-Prof. Priv.-Doz. Dr., Medical University of Vienna
Other Study IDs: VALID 1928/2017
Record Dates: First submitted 2018-05-06; First posted 2018-05-30 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Vascular Liver Disease; Portal Vein Thrombosis; Budd-Chiari Syndrome; Non-Cirrhotic Portal Hypertension; Rendu Osler Weber; Cardiac Cirrhosis; Porto-sinusoidal Vascular Disorder
MeSH Terms: conditions — Budd-Chiari Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — Blood, stool, urine, liver tissue, tissue from the lower / upper gastrointestinal tract (biopsy)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this Register Trial is to systematically study the epidemiology, risk factors, liver function as well prognosis of patients with vascular liver diseases. Furthermore, important clinical parameters will be assessed in order to evaluate patients' coagulation status and in order to develop new biomarkers derived from blood, urine, stool or ascites of patients as well as histological samples from the upper / lower GI-tract or the liver in order to better understand the natural history of vascular liver diseases.

DETAILED DESCRIPTION:
We will include patients with vascular liver diseases, including

* portal vein thrombosis (PVT)
* Budd-Chiari Syndrome (BCS)
* Heredetary Hemorrhagic Teleangiectasia (HHT, or Osler-Rendu Disease)
* Noncirrhotic-portal hypertension (NCPH) and Porto-sinusoidal vascular disorder
* Cirrhosis cardiaque if the fulfill inclusion/exclusion criteria and provide written informed consent. Participation in the biobank is optional for the patients. In particular, we will study the natural course of the patients in regard to hepatic decompensation (ascites, variceal bleeding, hepatic encephalopathy), need for intensified treatment (TIPS, ICU, liver transplantation) and survival.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a vascular liver disease by imaging (sonography, CT, MRI), transient elastography or liver histology
* PVT: Portal vein thrombosis
* NCPH: non-cirrhotic Portal Hypertension
* PSVD: porto-sinusoidal vascular disorder
* BCS: Budd-Chiari-Syndrome
* SOS: sinusoidal occlusive disease
* HHT: hereditary hemorrhagic teleangiectasia
* CIRCAD: cirrhosis cardiaque
* Age >18 years and <100 years
* Written informed consent obtained

Exclusion Criteria:

- withdrawal of written informed consent

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All consecutive patients with a vascular liver disease (as specified above) presenting at the outpatient department / inpatient ward of the Medical University of Vienna.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-12-12 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Hepatic Decompensation | Up to 10 years (=Study Period)
  Any first hepatic decompensation: variceal bleeding, new onset of ascites, new onset of hepatic encephalopathy, new onset of jaundice

SECONDARY OUTCOMES:
Liver-related death | Up to 10 years (=Study Period)
  Death from a liver-related cause
Coagulation status | Up to 10 years (=Study Period)
  Coagulation status of the Patient as assessed by advanced coagulation tests (including TEG-ROTEM and TGA)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria